CLINICAL TRIAL: NCT01270659
Title: Fentanyl Administered Intraorally for Rapid Treatment of Orthopedic Pain: The FAIRTOP II Trial
Brief Title: Safety and Efficacy Study of Fentanyl Buccal Tablet Use in the Emergency Department for Isolated Extremity Injury
Acronym: FAIRTOP II
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 1774
Record Dates: First submitted 2011-01-04; First posted 2011-01-05 (Estimated); Results first posted 2017-06-20 (Actual); Last update posted 2017-06-20 (Actual); Status verified 2017-05

CONDITIONS: Pain
Keywords: Fentanyl buccal tablet
MeSH Terms: conditions — Pain | interventions — Fentanyl; oxycodone-acetaminophen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Low-FBT (Experimental): Subject will receive FBT and placebo at a low dose
  Interventions: Drug: Fentanyl
- High-FBT (Experimental): Subject will receive the high dose regimen of FBT and a high dose placebo
  Interventions: Drug: Fentanyl
- Low control (Active Comparator): Subject will receive active oxycodone/APAP 5/325 mg and lansoprazole solutab for the fentanyl "placebo"
  Interventions: Drug: Oxycodone/acetaminophen
- High control (Active Comparator): Subject will receive the higher dose of the active comparator, #2 oxycodone/APAP 5/325mg, and lansoprazole solutab for the fentanyl "placebo"
  Interventions: Drug: oxycodone/acetaminophen

INTERVENTIONS:
Drug: Fentanyl — Fentanyl buccal tablet 100 mcg once
  Other Names: Fentora 100 mcg buccal tablet
  Arms: Low-FBT
Drug: Fentanyl — Fentanyl buccal tablet 200 mcg once
  Other Names: Fentora buccal tablet 200 mcg
  Arms: High-FBT
Drug: Oxycodone/acetaminophen — Oxycodone/acetaminophen 5/325 mg once
  Other Names: Percocet 5/325
  Arms: Low control
Drug: oxycodone/acetaminophen — Oxycodone/acetaminophen tablet 5/325 mg, 2 tablets one time
  Other Names: Percocet 5/325
  Arms: High control

SUMMARY:
The primary purpose of this study is to evaluate fentanyl buccal tablet (FBT) for analgesia in comparison to standard analgesia, to determine if the FBT allows for faster achievement of "significant analgesia"

DETAILED DESCRIPTION:
The subjects/patients will be asked if they would desire a low dose or high dose pain medication regimen. The low dose (low-FBT) group will receive FBT at a dose of 100 mcg, as well as an oral (pill) placebo preparation. The low dose (low-control) group will receive an "inactive comparator" (lansoprazole rapidly-dissolving buccal 15mg, " FBT placebo") and a dose of 5/325 Percocet tablet (oxycodone/acetaminophen 5/325). The high dose (high-FBT) group will receive 200 mcg FBT plus 2 placebo tablets. The high dose (high-control) group will receive the "FBT placebo" and a dose of 2, 5/325 Percocet tablets.

ELIGIBILITY:
Inclusion Criteria:

* pain sufficient to warrant medication stronger than acetaminophen (Tylenol) or aspirin
* only if Emergency Department provider approves
* a negative pregnancy test is required for participation for women of childbearing age

Exclusion Criteria:

* If treating provider determines intravenous analgesia is required
* allergy to acetaminophen or any opiate/opioid, or lansoprazole patients currently taking phenothiazines, CNS depressants (including alcohol), or if they have taken an monoamine oxidase inhibitor (MAOI) or selective serotonin reuptake inhibitor (SSRI) in the past two weeks
* if patient has already been administered an opioid analgesic for their current injury
* patients on chronic opioids therapy or a history of opioid abuse
* breastfeeding mothers
* patients who plan to drive home after their emergency department visit
* history of phenylketonuria (due to phenylalanine in the formulation of the lansoprazole solutab)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2011-05; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen H Thomas, MD MPH, Principal Investigator — University of Oklahoma; Annette O Arthur, PharmD, Study Director — University of Oklahoma
Locations (1):
- Hillcrest Medical Center Emergency Department, Tulsa, Oklahoma, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Low-FBT | High-FBT | Low Control | High Control
Started | 6 | 25 | 4 | 25
Completed | 6 | 25 | 4 | 25
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low-FBT | High-FBT | Low Control | High Control | Total
Number analyzed (Participants) | 6 | 25 | 4 | 25 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 2 | 0 | 1 | 4
  Between 18 and 65 years | 5 | 23 | 4 | 24 | 56
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.5 (10.01) | 38.4 (13.7) | 34.0 (13.1) | 35.4 (11.9) | 35.6 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 9 | 2 | 13 | 26
  Male | 4 | 16 | 2 | 12 | 34
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: White | 4 | 14 | 3 | 17 | 38
  Race/Ethnicity: Black | 2 | 10 | 0 | 7 | 19
  Race/Ethnicity: American Indian | 0 | 0 | 1 | 1 | 2
  Race/Ethnicity: Hispanic | 0 | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 6 | 25 | 4 | 25 | 60

OUTCOME MEASURES:

1. Primary Outcome: Median Time to Significant Analgesia (at Least 2 Units Decrease in Pain Level)
Description: Median time (in minutes) to 2 units decrease in pain level after drug administration. Patients were asked to rate their pain at every 5 minutes intervals from 0 to 60 minutes post drug administration. The 10-point verbally administered numeric pain rating scale (NPRS) was used to have patients rate their level of pain on a scale of 0 (no pain) to 10 (worst pain ever).
Time Frame: 60 minutes
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | Low-FBT | High-FBT | Low Control | High Control
Number analyzed (Participants) | 6 | 25 | 4 | 25
minutes | 15.0 [5.0 to NA] — Due to small sample size not enough participants achieved response to calculate upper limit. | 20.0 [15.0 to 25.0] | 15.0 [5.0 to NA] — Due to small sample size not enough participants achieved response to calculate upper limit. | 15.0 [10.0 to 25.0]

2. Secondary Outcome: Nausea Level
Description: Subjects' nausea level was recorded to determine how fentanyl buccal tablet compares to standard therapy in causing nausea. Treatment induced nausea and severity of nausea level was assessed.
  Nausea was assessed by a 10-point verbally administered scale. Patients rated their degree of nausea on a scale of 0 (no nausea) to 10 (worst nausea).
  At the beginning of the study, literature review found relatively little evidence guiding objective means to rate nausea, but there was some precedent for this approach (Warden C. Prehospital use of ondansetron reduces nausea and episodes of vomiting in adults and children over 12 years old [abstract]. Prehosp Emerg Care. 2007;11:132).
Time Frame: every 5 minutes for the first 60 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Low-FBT | High-FBT | Low Control | High Control
Number analyzed (Participants) | 6 | 25 | 4 | 25
Participants | 0 | 0 | 0 | 0

3. Secondary Outcome: Number of Participants Experiencing Any Adverse Events
Description: Occurrence of any adverse event.
Time Frame: Full 2 hours of the study period
Measure: Count of Participants; unit: Participants
Arm/Group | Low-FBT | High-FBT | Low Control | High Control
Number analyzed (Participants) | 6 | 25 | 4 | 25
Participants | 1 | 9 | 3 | 10

ADVERSE EVENTS:
Time Frame: All study patients were monitored during the entire study period i.e., 2 hours after medication administration.
Arm/Group | Low-FBT | High-FBT | Low Control | High Control
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/25 | 0/4 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/25 | 0/4 | 0/25
Other Adverse Events (participants affected / at risk) | 1/6 | 9/25 | 3/4 | 10/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Low-FBT (N=6) | High-FBT (N=25) | Low Control (N=4) | High Control (N=25)
Nausea (Gastrointestinal disorders) | 0 | 3 | 0 | 5
Pruritis (Skin and subcutaneous tissue disorders) | 1 | 1 | 3 | 2
Headache (Nervous system disorders) | 0 | 0 | 0 | 4
Dry mouth (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Drowsy (Nervous system disorders) | 0 | 4 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes